CLINICAL TRIAL: NCT01572129
Title: Clopidogrel Reloading in Patients With Non-ST Elevation Acute Coronary Syndrome Undergoing PCI on Chronic Clopidogrel Therapy. Results of the ARMYDA RELOAD ACS (Antiplatelet Therapy for Reduction of MYocardial Damage During Angioplasty in Acute Coronary Syndrome) Randomized Trial.
Brief Title: Clopidogrel Reloading in Patients With NSTEACS Undergoing Percutaneous Coronary Intervention on Chronic Clopidogrel Therapy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Campus Bio-Medico University (Other)
Responsible Party: Principal Investigator, Patti Giuseppe, MD, FACC, Co-Chair of the ARMYDA Study Group, Assistant Professor of Cardiology, Campus Bio-Medico University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2011-005449-11
Record Dates: First submitted 2012-04-03; First posted 2012-04-06 (Estimated); Last update posted 2012-04-06 (Estimated); Status verified 2012-04

CONDITIONS: Acute Coronary Syndrome; Myocardial Infarction
MeSH Terms: conditions — Acute Coronary Syndrome; Myocardial Infarction | interventions — Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Reload (Experimental): 600 mg of clopidogrel loading dose 6-8 h before coronary angiogram, in addition to the chronic daily dose of 75 mg
  Interventions: Drug: Clopidogrel
- Placebo (Placebo Comparator): Placebo arm in addition to the chronic daily dose of 75 mg
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Clopidogrel — 600 mg clopidogrel loading dose 6-8 h before diagnostic coronary angiogram
  Other Names: Plavix
  Arms: Reload
Drug: Placebo — Placebo in addition to the chronic daily dose of 75 mg
  Arms: Placebo

SUMMARY:
Patients who developed an acute coronary syndrome despite dual antiplatelet therapy with aspirin and clopidogrel may benefit from a further dose of clopidogrel before a percutaneous coronary intervention.

The aim of this study is to evaluate safety and effectiveness of clopidogrel reloading in patients on chronic clopidogrel therapy with acute coronary syndrome undergoing percutaneous coronary intervention.

ELIGIBILITY:
Inclusion Criteria:

* chronic (> 10 days) therapy with clopidogrel (75 mg/day)
* non-ST-segment elevation acute coronary syndrome (ACS) requiring early diagnostic angiography

Exclusion Criteria:

* primary percutaneous coronary intervention (PCI) for acute ST-segment elevation acute myocardial infarction
* platelet count < 70 × 10^9/L
* high bleeding risk
* coronary bypass grafting in the previous 3 months

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2011-11; Primary Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiovascular Events | 30 days
  Death Myocardial Infarction Target Vessel Revascularization

SECONDARY OUTCOMES:
Bleeding Events | 30 days
  Occurrence of vascular/bleeding complications, defined as: (a) major bleeding (intracranial bleeding or clinically overt bleeding associated with a decrease in haemoglobin >5 g/dL, according to the TIMI criteria); (b) minor bleeding (clinically overt haemorrhage associated with a fall in haemoglobin ≤5 g/dL); (c) entry-site complications (haematoma >5 cm, pseudoaneurysm or arteriovenous fistula)
Grade of platelet residual reactivity | Immediately before PCI (4-6h after randomization), 8h and 24h after PCI
  Patient's response to clopidogrel at 3 different timing, assessed with VerifyNow P2Y12 Assays.
  The first timing is immediately before PCI (4-6h after randomization), once accomplished the diagnostic angiogram.
  The second and third timings are, respectively, 8h and 24h after PCI.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Patti, MD, Principal Investigator — Campus Bio-Medico University
Locations (2):
- Italy (2):
  - Vito Fazzi Hospital, Lecce, Lecce
  - Campus Bio-Medico University, Rome, Rome

REFERENCES:
- [Background] Di Sciascio G, Patti G, Pasceri V, Colonna G, Mangiacapra F, Montinaro A; ARMYDA-4 RELOAD Investigators. Clopidogrel reloading in patients undergoing percutaneous coronary intervention on chronic clopidogrel therapy: results of the ARMYDA-4 RELOAD (Antiplatelet therapy for Reduction of MYocardial Damage during Angioplasty) randomized trial. Eur Heart J. 2010 Jun;31(11):1337-43. doi: 10.1093/eurheartj/ehq081. Epub 2010 Apr 2. PMID 20363764
- [Background] Kastrati A, von Beckerath N, Joost A, Pogatsa-Murray G, Gorchakova O, Schomig A. Loading with 600 mg clopidogrel in patients with coronary artery disease with and without chronic clopidogrel therapy. Circulation. 2004 Oct 5;110(14):1916-9. doi: 10.1161/01.CIR.0000137972.74120.12. Epub 2004 Jul 19. PMID 15262828